CLINICAL TRIAL: NCT00545714
Title: Multicentre, Non-Randomised, Open-Label Phase II Study to Evaluate the Efficacy and Safety of Induction Treatment With Rituximab, Fludarabine, Cyclophosphamide, Followed by Rituximab Maintenance Therapy (R-Fc-Rm) in the First Line Treatment of Chronic Lymphocytic Leukaemia
Brief Title: A Study to Assess the Efficacy of Rituximab (MabThera) in First Line Treatment of Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21135; 2007-002733-36 (EudraCT Number)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine; Rituximab

ARMS (1):
- Rituximab + Fludarabine + Cyclophosphamide (Experimental): Participants will receive 6 cycles (cycle length = 28 days) of treatment with rituximab (375 milligrams per square meter [mg/m^2] as intravenous [IV] infusion on Day 0 of Cycle 1 and 500 mg/m^2 as IV infusion on Day 1 of Cycles 2-6); fludarabine (25 mg/m^2 on Days 1-3) and cyclophosphamide (250 mg/m^2 on Days 1-3). Participants with a partial or complete response and appropriate neutrophil conditions will receive maintenance treatment with rituximab (375 mg/m^2 as IV infusion every 2 months) from 3 months after Day 1 Cycle 6 up to a total of 18 doses or up to 3 years after Cycle 6.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 250 mg/m^2 as IV infusion will be administered on Days 1-3 of first six 28-day cycles.
Drug: Fludarabine — Fludarabine 25 mg/m^2 as IV infusion will be administered on Days 1-3 of first six 28-day cycles.
Drug: Rituximab — Rituximab 375 mg/m^2 as IV infusion will be administered on Day 0 of Cycle 1; 500 mg/m^2 as IV infusion will be administered on Day 1 of Cycle 2-6; and 375 mg/m^2 as IV infusion every 2 months from 3 months after Day 1 Cycle 6 up to a total of 18 doses or up to 3 years after Cycle 6.
  Other Names: MabThera, Rituxan

SUMMARY:
This single arm study will assess the efficacy and safety of rituximab in combination with fludarabine and cyclophosphamide, followed by rituximab maintenance therapy, as first line treatment of participants with CLL.

ELIGIBILITY:
Inclusion Criteria:

* CLL according to World Health Organization diagnostic criteria
* Active disease
* No previous treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Exclusion Criteria:

* Transformation to aggressive B-cell malignancy (prolymphocytic leukemia, large-cell lymphoma, Hodgkin's lymphoma)
* Other malignancies except for localized skin cancer
* Continuous systemic corticosteroid treatment
* Known infection with hepatitis B or C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-11-21 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Spain (33):
  - Hospital De Txagorritxu; Servicio de Hematologia, Vitoria-Gasteiz, Alava
  - Hospital Universitario Puerta del Mar; Servicio de Hematologia, Cadiz, Cadiz
  - Hospital de Jerez de la Frontera; Servicio de Hematologia, Jerez de la Frontera, Cadiz
  - Hospital Universitario Marques de Valdecilla; Servicio de Hematologia, Santander, Cantabria
  - Hospital General de Castellon; Servicio de Hematologia, Castellon, Castellon
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Hematologia, A Coruña, LA Coruña
  - Fundacion Hospital de Alcorcon; Servicio de Hematologia, Alcorcón, Madrid
  - Hosital Universitario de Mostoles;Servicio de Hematologia, Móstoles, Madrid
  - Hospital Francesc de Borja; Servicio de Hematologia, Gandia, Valencia
  - Hospital de Sagunto; Servicio de Hematologia, Sagunto, Valencia
  - Hospital de Basurto; Servicio de Hematologia, Bilbao, Vizcaya
  - Hospital Universitario Infanta Cristina; Servicio de Hematologia, Badajoz
  - Hospital Duran i Reynals; Servicio de Hematologia, Barcelona
  - Hospital San Pedro De Alcantara; Servicio de Hematologia, Cáceres
  - Hospital Universitario Virgen de las Nieves; Servicio de Hematologia, Granada
  - Hospital General Universitario Gregorio Marañon; Servicio de Hematología, Madrid
  - Hospital Ramon y Cajal; Servicio de Hematologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Hematología, Madrid
  - Hospital Univ. 12 de Octubre; Servicio de Hematologia, Madrid
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio Hematologia, Madrid
  - Hospital Universitario Puerta de Hierro; Servicio de Hematologia, Madrid
  - Hospital Universitario Principe de Asturias; Servicio de Hematología, Madrid
  - Hospital Universitario de Getafe; Servico de Hematologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Hematologia, Málaga
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Hematología, Murcia
  - Hospital Clinico Universitario de Salamanca;Servicio de Hematologia, Salamanca
  - Hospital General Universitario de Valencia; Servicio de Hematologia, Valencia
  - Hospital Arnau de Vilanova (Valencia) Servicio de Hematologia, Valencia
  - Hospital Universitario Dr. Peset; Servicio de Hematologia, Valencia
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Hematologia, Zaragoza
  - Hospital Universitario Miguel Servet; Servicio Hematologia, Zaragoza

REFERENCES:
- [Derived] Garcia-Marco JA, Jimenez JL, Recasens V, Zarzoso MF, Gonzalez-Barca E, De Marcos NS, Ramirez MJ, Parraga FJP, Yanez L, De La Serna Torroba J, Malo MDG, Ariznavarreta GD, Persona EP, Guinaldo MAR, De Paz Arias R, Llanos EB, Jarque I, Valle MDCF, Tatay AC, De Oteyza JP, Martin EMD, Fernandez IP, Martinez RM, Costa MAA, Champ D, Suarez JG, Diaz MG, Ferrer S, Carbonell F, Garcia-Vela JA; GELLC Study Group. High prognostic value of measurable residual disease detection by flow cytometry in chronic lymphocytic leukemia patients treated with front-line fludarabine, cyclophosphamide, and rituximab, followed by three years of rituximab maintenance. Haematologica. 2019 Nov;104(11):2249-2257. doi: 10.3324/haematol.2018.204891. Epub 2019 Mar 19. PMID 30890600

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 86 participants were enrolled in 29 centers in Spain in this two-phase study (Induction Phase and Maintenance Phase).
Groups:
- Rituximab + Fludarabine + Cyclophosphamide: Participants received rituximab 375 milligrams per square meter (mg/m^2) as intravenous (IV) infusion on Day 0 of Cycle 1 and 500 mg/m^2 as IV infusion on Day 1 of Cycles 2-6 (cycle length = 28 days); fludarabine 25 mg/m^2 on Days 1-3 of each cycle and cyclophosphamide 250 mg/m^2 on Days 1-3 of each cycle during the Induction Phase. Participants with a partial response (PR) or complete response (CR) and appropriate neutrophil conditions received maintenance treatment with rituximab (375 mg/m^2 as IV infusion every 2 months) from 3 months after Day 1 Cycle 6 up to a total of 18 doses or up to 3 years after Cycle 6 of Induction Phase.
Period: Induction Phase (6 Months)
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Started | 86
Safety Population | 86
Intent-to-Treat (ITT) Population | 84
Completed | 74
Not Completed | 12
Not completed — Physician Decision | 3
Not completed — Unacceptable Toxicity | 6
Not completed — Disease Progression | 1
Not completed — Eligibility Criteria Violation | 2
Period: Maintenance Phase (36 Months)
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Started | 74
Completed | 42
Not Completed | 32
Not completed — Unacceptable Toxicity | 16
Not completed — Disease Progression | 9
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all participants who received at least one dose of study drug and met inclusion/exclusion criteria.
Groups:
- Rituximab + Fludarabine + Cyclophosphamide: Participants received rituximab 375 mg/m^2 as IV infusion on Day 0 of Cycle 1 and 500 mg/m^2 as IV infusion on Day 1 of Cycles 2-6 (cycle length = 28 days); fludarabine 25 mg/m^2 on Days 1-3 of each cycle and cyclophosphamide 250 mg/m^2 on Days 1-3 of each cycle during the Induction Phase. Participants with a PR or CR and appropriate neutrophil conditions received maintenance treatment with rituximab (375 mg/m^2 as IV infusion every 2 months) from 3 months after Day 1 Cycle 6 up to a total of 18 doses or up to 3 years after Cycle 6 of Induction Phase.
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.92 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With CR Achieved After the Rituximab, Fludarabine, and Cyclophosphamide Regimen
Description: CR was defined as no adenopathies (ADPs) and visceromegalies (VSMs) in physical examination (PE); no general symptoms (Sx); lymphocytes (Lymph) in peripheral blood less than (<) 4000 per cubic millimeter (mm^3); normalization of peripheral blood parameters: neutrophils (Neut) greater than (>) 1500/mm^3, platelets (Plt) >100,000/mm^3, hemoglobin (Hb) >11 grams per deciliter (g/dL) without transfusion; normocellular bone marrow (BM) with <30% Lymph; BM aspirate/biopsy with no evidence of infiltration of lymphoid nodules.
Time Frame: Month 9
Population: ITT Population included all participants who received at least one dose of study drug and met inclusion/exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Percentage of Participants | 95.2 [88.25 to 98.69]

2. Secondary Outcome: Percentage of Participants With Clinical Response of CR or PR as Assessed by Multiparameter Flow Cytometry
Description: CR was defined as no ADPs and VSMs in PE; no general Sx; Lymph in peripheral blood <4000/mm^3; normalization of peripheral blood parameters: Neut >1500/mm^3, Plt >100,000/mm^3, Hb >11 g/dL without transfusion; normocellular BM with <30% Lymph; BM aspirate/biopsy with no evidence of infiltration of lymphoid nodules. PR was defined as decrease >50% in Lymph in peripheral blood; reduction in ADPs >50% in total sum of up to 6 ADPs or in the baseline ADP of largest diameter (LD), no new ADP or enlargement of a prior ADP; >50% decrease in VSM; Neut >1500/mm^3 or >50% increase from Baseline; Plt >100,000/mm^3 or >50% increase from Baseline; Hb >11.0 g/dL or >50% increase from Baseline value without transfusion. Participants who met all CR criteria but had persistent anemia or thrombocytopenia were considered as PR.
Time Frame: Post-Induction Phase (IP): at 6 months; during Maintenance Phase (MP): at Cycles 9, 12, 15, 18 (cycle length = 2 months); during Follow-Up (FU): at Follow-Up Months 6, 12, 18, 24, 30, 36
Population: ITT Population. Here, 'Number Analyzed' signifies participants who were evaluable for indicated category.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Percentage of Participants
  Post-IP: CR | 75.0
  Post-IP: PR | 13.1
  MP (9 Cycles): CR: number analyzed (Participants) | 47
  MP (9 Cycles): CR | 89.4
  MP (9 Cycles): PR: number analyzed (Participants) | 47
  MP (9 Cycles): PR | 6.4
  MP (12 Cycles): CR: number analyzed (Participants) | 33
  MP (12 Cycles): CR | 87.9
  MP (12 Cycles): PR: number analyzed (Participants) | 33
  MP (12 Cycles): PR | 6.1
  MP (15 Cycles): CR: number analyzed (Participants) | 22
  MP (15 Cycles): CR | 90.9
  MP (15 Cycles): PR: number analyzed (Participants) | 22
  MP (15 Cycles): PR | 4.5
  MP (18 Cycles): CR: number analyzed (Participants) | 59
  MP (18 Cycles): CR | 88.1
  MP (18 Cycles): PR: number analyzed (Participants) | 59
  MP (18 Cycles): PR | 8.5
  6 Months FU: CR: number analyzed (Participants) | 12
  6 Months FU: CR | 83.3
  6 Months FU: PR: number analyzed (Participants) | 12
  6 Months FU: PR | 0.0
  12 Months FU: CR: number analyzed (Participants) | 36
  12 Months FU: CR | 94.4
  12 Months FU: PR: number analyzed (Participants) | 36
  12 Months FU: PR | 0.0
  18 Months FU: CR: number analyzed (Participants) | 2
  18 Months FU: CR | 100.0
  18 Months FU: PR: number analyzed (Participants) | 2
  18 Months FU: PR | 0.0
  24 Months FU: CR: number analyzed (Participants) | 29
  24 Months FU: CR | 93.1
  24 Months FU: PR: number analyzed (Participants) | 29
  24 Months FU: PR | 0.0
  30 Months FU: CR: number analyzed (Participants) | 2
  30 Months FU: CR | 100.0
  30 Months FU: PR: number analyzed (Participants) | 2
  30 Months FU: PR | 0.0
  36 Months FU: CR: number analyzed (Participants) | 31
  36 Months FU: CR | 100.0
  36 Months FU: PR: number analyzed (Participants) | 31
  36 Months FU: PR | 0.0

3. Secondary Outcome: Percentage of Participants With Clinical Response of CR or PR Among Participants With Negative Minimal Residual Disease (MRD) as Assessed by Multiparameter Flow Cytometry
Description: CR: no ADPs and VSMs in PE; no general Sx; Lymph in peripheral blood <4000/mm^3; normalization of peripheral blood parameters: Neut >1500/mm^3, Plt >100,000/mm^3, Hb >11 g/dL without transfusion; normocellular BM with <30% Lymph; BM aspirate/biopsy with no evidence of infiltration of lymphoid nodules. PR: decrease >50% in Lymph in peripheral blood; reduction in ADPs >50% in total sum of up to 6 ADPs or in the baseline ADP of largest diameter (LD), no new ADP or enlargement of a prior ADP; >50% decrease in VSM; Neut >1500/mm^3 or >50% increase from Baseline; Plt >100,000/mm^3 or >50% increase from Baseline; Hb >11.0 g/dL or >50% increase from Baseline value without transfusion. Participants who met all CR criteria but had persistent anemia or thrombocytopenia were considered as PR. Negative MRD: Lymph <0.01% of all white blood cells (WBCs) in blood or BM after two consecutive measurements. Analysis performed only in blood during the Maintenance Phase and Follow-Up.
Time Frame: Post-Induction Phase: at 6 months; during Maintenance Phase: at Cycles 9, 12, 15, 18 (cycle length = 2 months); during Follow-Up: at Follow-Up Months 6, 12, 18, 24, 36
Population: ITT Population. Only those with negative MRD were included in the analysis. Here, 'Number Analyzed' signifies participants who were evaluable for indicated category.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 60
Percentage of Participants
  Post-IP: Blood MRD Negative | 100.0
  Post-IP: BM MRD Negative: number analyzed (Participants) | 37
  Post-IP: BM MRD Negative | 100.0
  MP (9 Cycles): Blood MRD Negative: number analyzed (Participants) | 33
  MP (9 Cycles): Blood MRD Negative | 100.0
  MP (12 Cycles): Blood MRD Negative: number analyzed (Participants) | 22
  MP (12 Cycles): Blood MRD Negative | 100.0
  MP (15 Cycles): Blood MRD Negative: number analyzed (Participants) | 16
  MP (15 Cycles): Blood MRD Negative | 100.0
  MP (18 Cycles): Blood MRD Negative: number analyzed (Participants) | 40
  MP (18 Cycles): Blood MRD Negative | 100.0
  6 Months FU: Blood MRD Negative: number analyzed (Participants) | 4
  6 Months FU: Blood MRD Negative | 100.0
  12 Months FU: Blood MRD Negative: number analyzed (Participants) | 24
  12 Months FU: Blood MRD Negative | 100.0
  18 Months FU: Blood MRD Negative: number analyzed (Participants) | 1
  18 Months FU: Blood MRD Negative | 100.0
  24 Months FU: Blood MRD Negative: number analyzed (Participants) | 19
  24 Months FU: Blood MRD Negative | 100.0
  36 Months FU: Blood MRD Negative: number analyzed (Participants) | 22
  36 Months FU: Blood MRD Negative | 100.0

4. Secondary Outcome: Percentage of Participants With CR With Incomplete Bone Marrow Recovery (CRi)
Description: Participants with CRi were those who met all CR criteria (including BM examinations) but had persistent anemia, thrombocytopenia, or neutropenia apparently unrelated to chronic lymphocytic leukemia (CLL) but related to drug toxicity. CR: no ADPs and VSMs in PE; no general Sx; Lymph in peripheral blood <4000/mm^3; normalization of peripheral blood parameters: Neut >1500/mm^3, Plt >100,000/mm^3, Hb >11 g/dL without transfusion; normocellular BM with <30% Lymph; BM aspirate/biopsy with no evidence of infiltration of lymphoid nodules.
Time Frame: Baseline up to progressive disease (PD) or death due to any cause, whichever occurred first (up to 92 months)
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Percentage of Participants | 7.1

5. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Baseline up to death due to any cause (up to 92 months)
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 86
Percentage of Participants | 23.2 [5.72 to NA]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from treatment start to death of the participant. For all other participants, the last follow-up available was taken as the last control. If the participant had not completed the study, the date of the last visit available was considered. OS was estimated using Kaplan-Meier (KM) methodology.
Time Frame: Baseline up to death due to any cause (up to 92 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Years | 7.51 [7.5 to NA] — The upper limit of confidence interval (CI) was not estimable due to high number of censored participants.

7. Secondary Outcome: Percentage of Participants With PD or Death
Description: PD was defined as new ADPs (1.5 centimeters [cm]), hepato-/splenomegaly (HSM), Richter syndrome (RS), or other infiltrated organs; greater than or equal to (>/=) 50% increase in size of Baseline prior ADPs or HSM in participants with PR; Lymph increase >/=50% in peripheral blood with B Lymph >/=5000/mm^3; cytopenia attributable to CLL. Progression of any cytopenia (not related to autoimmune cytopenia) reported as a 2-g/dL decrease in basal Hb, Hb <10 g/dL, >/=50% decrease in basal Plt count, or count <100,000/mm^3 at >/=3 months post-treatment was defined as PD if BM biopsy confirmed infiltration of clonal CLL cells.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to 92 months)
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Percentage of Participants | 39.29 [5.72 to NA]

8. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from start of study treatment to PD or death, whichever occurred first. For other participants, last follow-up available was taken as last control. If participant did not complete study, date of last visit available was considered. PFS was estimated using KM methodology. PD was defined as new ADPs (1.5 cm), HSM, RS, or other infiltrated organs; >/=50% increase in size of Baseline prior ADPs or HSM in participants with PR; Lymph increase >/=50% in peripheral blood with B Lymph >/=5000/mm^3; cytopenia attributable to CLL. Progression of any cytopenia (not related to autoimmune cytopenia) reported as a 2-g/dL decrease in basal Hb, Hb <10 g/dL, >/=50% decrease in basal Plt count, or count <100,000/mm^3 at >/=3 months post-treatment was defined as PD if BM biopsy confirmed infiltration of clonal CLL cells.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to 92 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Years | 6.96 [5.72 to NA] — The upper limit of CI was not estimable due to high number of censored participants.

9. Secondary Outcome: Treatment-Free Survival (TFS)
Description: TFS was defined time from start of study treatment until participant received new chemotherapy/immunotherapy because of PD and to reduce the disease with palliative or curative intent. PD was defined as new ADPs (1.5 cm), HSM, RS, or other infiltrated organs; >/=50% increase in size of Baseline prior ADPs or HSM in participants with PR; Lymph increase >/=50% in peripheral blood with B Lymph >/=5000/mm^3; cytopenia attributable to CLL. Progression of any cytopenia (not related to autoimmune cytopenia) reported as a 2-g/dL decrease in basal Hb, Hb <10 g/dL, >/=50% decrease in basal Plt count, or count <100,000/mm^3 at >/=3 months post-treatment was defined as PD if BM biopsy confirmed infiltration of clonal CLL cells.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to 92 months)
Population: ITT Population. Only those who received new chemotherapy/immunotherapy, as per definitions for TFS, were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 27
Years | 4.13 [2.98 to 4.87]

10. Secondary Outcome: Duration of Response (DOR)
Description: DOR: time from CR/PR to MRD/PD. PD: new ADP (1.5 cm), HSM, RS, other infiltrated organs or >/=50% increase size in those with PR; blood Lymph increase >/=50% with B Lymph >/=5000/mm^3; cytopenia due to CLL. Progression of (nonautoimmune) cytopenia: 2-g/dL decrease basal Hb, Hb <10 g/dL, >/=50% decrease basal Plt or <100,000/mm^3 at >/=3 months post-treatment was PD if clonal CLL cell infiltration on BM biopsy. CR: no ADP/VSM in PE; no general Sx; blood Lymph <4000/mm^3; Neut >1500/mm^3; Plt >100,000/mm^3; Hb >11 g/dL (no transfusion); normocellular BM with <30% Lymph; BM aspirate/biopsy with no lymphoid nodule infiltration. PR: >50% decrease blood Lymph; >50% decrease in total sum up to 6 ADPs or baseline ADP of LD, no new/enlargement of prior ADP; >50% decrease VSM; Neut >1500/mm^3 or >50% increase; Plt >100,000/mm^3 or >50% increase; Hb >11.0 g/dL or >50% increase (no transfusion). All CR criteria but persistent anemia or thrombocytopenia was PR. MRD: Lymph >0.01% of blood/BM WBCs.
Time Frame: From first CR or PR up to detectable MRD or disease occurrence/PD, whichever occurred first (up to 92 months)
Population: ITT Population. Only those participants who achieved a clinical response of CR or PR were evaluable for this measure.
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 80
Years | NA [NA to NA] — Median time of response was not estimable due to high number of censored participants.

11. Secondary Outcome: Percentage of Participants With Cluster of Differentiation (CD) 38 Cells >/=30% in Peripheral Blood
Description: Percentages of participants with CD38 expression by >/=30% of CLL cells during the Induction Phase, Maintenance Phase, and Follow-Up were reported.
Time Frame: Post-Induction Phase: at 6 months; during Maintenance Phase: at Cycles 9, 12, 15, 18 (cycle length = 2 months); during Follow-Up: at Follow-Up Months 6, 12, 18, 24, 30, 36
Population: ITT Population. Here, 'Number Analyzed' signifies participants who were evaluable for indicated category.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Percentage of Participants
  Post-IP | 47.6
  MP (9 Cycles): number analyzed (Participants) | 47
  MP (9 Cycles) | 44.4
  MP (12 Cycles): number analyzed (Participants) | 33
  MP (12 Cycles) | 45.5
  MP (15 Cycles): number analyzed (Participants) | 22
  MP (15 Cycles) | 47.6
  MP (18 Cycles): number analyzed (Participants) | 59
  MP (18 Cycles) | 47.4
  6 Months FU: number analyzed (Participants) | 12
  6 Months FU | 66.7
  12 Months FU: number analyzed (Participants) | 36
  12 Months FU | 45.7
  18 Months FU: number analyzed (Participants) | 2
  18 Months FU | 100.0
  24 Months FU: number analyzed (Participants) | 29
  24 Months FU | 41.4
  30 Months FU: number analyzed (Participants) | 2
  30 Months FU | 50.0
  36 Months FU: number analyzed (Participants) | 31
  36 Months FU | 35.5

12. Secondary Outcome: Percentage of Participants With Genetic Abnormalities
Description: Percentages of participants with genetic abnormalities (deletion 6q, deletion 11q22-q23, deletion p53, trisomy 12, and deletion 13q14) in the course of the disease during the Induction Phase and Maintenance Phase were reported.
Time Frame: Post-Induction Phase: at 6 months; during Maintenance Phase: at Cycles 9, 12, 15, 18 (cycle length = 2 months)
Population: ITT Population. Here, 'Number Analyzed' signifies participants who were evaluable for indicated category. Designation of 'MP (xC)' refers to number of cycles in Maintenance Phase.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Percentage of Participants
  Post-IP: Deletion 6q | 3.6
  Post-IP: Deletion 11q22-q23 | 26.2
  Post-IP: Deletion p53 | 4.8
  Post-IP: Trisomy 12 | 15.5
  Post-IP: Deletion 13q14 | 50.0
  MP (9C): Deletion 6q: number analyzed (Participants) | 47
  MP (9C): Deletion 6q | 4.3
  MP (9C): Deletion 11q22-q23: number analyzed (Participants) | 47
  MP (9C): Deletion 11q22-q23 | 25.5
  MP (9C): Deletion p53: number analyzed (Participants) | 47
  MP (9C): Deletion p53 | 0.0
  MP (9C): Trisomy 12: number analyzed (Participants) | 47
  MP (9C): Trisomy 12 | 17.0
  MP (9C): Deletion 13q14: number analyzed (Participants) | 47
  MP (9C): Deletion 13q14 | 55.3
  MP (12C): Deletion 6q: number analyzed (Participants) | 33
  MP (12C): Deletion 6q | 3.0
  MP (12C): Deletion 11q22-q23: number analyzed (Participants) | 33
  MP (12C): Deletion 11q22-q23 | 21.2
  MP (12C): Deletion p53: number analyzed (Participants) | 33
  MP (12C): Deletion p53 | 0.0
  MP (12C): Trisomy 12 (n= 33): number analyzed (Participants) | 33
  MP (12C): Trisomy 12 (n= 33) | 21.2
  MP (12C): Deletion 13q14: number analyzed (Participants) | 33
  MP (12C): Deletion 13q14 | 51.5
  MP (15C): Deletion 6q: number analyzed (Participants) | 22
  MP (15C): Deletion 6q | 4.5
  MP (15C): Deletion 11q22-q23: number analyzed (Participants) | 22
  MP (15C): Deletion 11q22-q23 | 31.8
  MP (15C): Deletion p53: number analyzed (Participants) | 22
  MP (15C): Deletion p53 | 0.0
  MP (15C): Trisomy 12: number analyzed (Participants) | 22
  MP (15C): Trisomy 12 | 18.2
  MP (15C): Deletion 13q14: number analyzed (Participants) | 22
  MP (15C): Deletion 13q14 | 59.1
  MP (18C): Deletion 6q: number analyzed (Participants) | 59
  MP (18C): Deletion 6q | 3.4
  MP (18C): Deletion 11q22-q23: number analyzed (Participants) | 59
  MP (18C): Deletion 11q22-q23 | 23.7
  MP (18C): Deletion p53: number analyzed (Participants) | 59
  MP (18C): Deletion p53 | 0.0
  MP (18C): Trisomy 12: number analyzed (Participants) | 59
  MP (18C): Trisomy 12 | 18.6
  MP (18C): Deletion 13q14: number analyzed (Participants) | 59
  MP (18C): Deletion 13q14 | 49.2

13. Secondary Outcome: Percentage of Participants With Positive and Negative Zeta-Chain-Associated Protein Kinase 70 (ZAP-70) Expression
Description: Percentages of participants with positive and negative ZAP-70 expression during the Induction Phase, Maintenance Phase, and Follow-Up were reported. Positive ZAP-70 was defined as ZAP-70 expression by >/=20% of CLL cells. Negative ZAP-70 was defined as ZAP-70 expression by <20% of CLL cells.
Time Frame: as for outcome 11
Population: ITT Population. Here, 'Number Analyzed' signifies participants who were evaluable for indicated category.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Percentage of Participants
  Post-IP: Positive | 57.3
  Post-IP: Negative | 42.7
  MP (9 Cycles): Positive: number analyzed (Participants) | 47
  MP (9 Cycles): Positive | 57.5
  MP (9 Cycles): Negative: number analyzed (Participants) | 47
  MP (9 Cycles): Negative | 42.5
  MP (12 Cycles): Positive: number analyzed (Participants) | 33
  MP (12 Cycles): Positive | 62.1
  MP (12 Cycles): Negative: number analyzed (Participants) | 33
  MP (12 Cycles): Negative | 37.9
  MP (15 Cycles): Positive: number analyzed (Participants) | 22
  MP (15 Cycles): Positive | 57.1
  MP (15 Cycles): Negative: number analyzed (Participants) | 22
  MP (15 Cycles): Negative | 42.9
  MP (18 Cycles): Positive: number analyzed (Participants) | 59
  MP (18 Cycles): Positive | 54.9
  MP (18 Cycles): Negative: number analyzed (Participants) | 59
  MP (18 Cycles): Negative | 45.1
  6 Months FU: Positive: number analyzed (Participants) | 12
  6 Months FU: Positive | 63.6
  6 Months FU: Negative: number analyzed (Participants) | 12
  6 Months FU: Negative | 36.4
  12 Months FU: Positive: number analyzed (Participants) | 36
  12 Months FU: Positive | 60.0
  12 Months FU: Negative: number analyzed (Participants) | 36
  12 Months FU: Negative | 40.0
  18 Months FU: Positive: number analyzed (Participants) | 2
  18 Months FU: Positive | 100.0
  18 Months FU: Negative: number analyzed (Participants) | 2
  18 Months FU: Negative | 0.0
  24 Months FU: Positive: number analyzed (Participants) | 29
  24 Months FU: Positive | 59.3
  24 Months FU: Negative: number analyzed (Participants) | 29
  24 Months FU: Negative | 40.7
  30 Months FU: Positive: number analyzed (Participants) | 2
  30 Months FU: Positive | 100.0
  30 Months FU: Negative: number analyzed (Participants) | 2
  30 Months FU: Negative | 0.0
  36 Months FU: Positive: number analyzed (Participants) | 31
  36 Months FU: Positive | 57.1
  36 Months FU: Negative: number analyzed (Participants) | 31
  36 Months FU: Negative | 42.9

14. Secondary Outcome: Percentage of Participants With Immunoglobulin Heavy Locus (IgH) Rearrangement
Description: Percentages of participants with IgH rearrangement during the Induction Phase, Maintenance Phase, and Follow-Up were reported.
Time Frame: as for outcome 11
Population: ITT Population. Here, 'Number Analyzed' signifies participants who were evaluable for indicated category.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 84
Percentage of Participants
  Post-IP | 36.2
  MP (9 Cycles): number analyzed (Participants) | 47
  MP (9 Cycles) | 37.1
  MP (12 Cycles): number analyzed (Participants) | 33
  MP (12 Cycles) | 20.0
  MP (15 Cycles): number analyzed (Participants) | 22
  MP (15 Cycles) | 29.4
  MP (18 Cycles): number analyzed (Participants) | 59
  MP (18 Cycles) | 33.3
  6 Months FU: number analyzed (Participants) | 12
  6 Months FU | 100.0
  12 Months FU: number analyzed (Participants) | 36
  12 Months FU | 37.9
  18 Months FU: number analyzed (Participants) | 2
  18 Months FU | 50.0
  24 Months FU: number analyzed (Participants) | 29
  24 Months FU | 33.3
  30 Months FU: number analyzed (Participants) | 2
  30 Months FU | 0.0
  36 Months FU: number analyzed (Participants) | 31
  36 Months FU | 45.8

ADVERSE EVENTS:
Time Frame: Baseline through end of Follow-Up (up to 92 months)
Description: Safety Population included all participants who received at least one dose of study drug.
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 35/86
Other Adverse Events (participants affected / at risk) | 82/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Fludarabine + Cyclophosphamide (N=86)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Malabsorption (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 6
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic mass (Hepatobiliary disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Meningitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Viral myocarditis (Infections and infestations) | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1
Vertebroplasty (Surgical and medical procedures) | 1
Capillary leak syndrome (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Fludarabine + Cyclophosphamide (N=86)
Leukopenia (Blood and lymphatic system disorders) | 15
Lymphopenia (Blood and lymphatic system disorders) | 24
Neutropenia (Blood and lymphatic system disorders) | 52
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 26
Vomiting (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 14
Chills (General disorders) | 6
Pyrexia (General disorders) | 31
Nasopharyngitis (Infections and infestations) | 27
Pneumonia (Infections and infestations) | 7
Respiratory tract infection (Infections and infestations) | 14
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/ or the publication be postponed in order to protect the Sponsor's intellectual property rights.